CLINICAL TRIAL: NCT05789407
Title: Is Exposure to Persistent Organic Pollutants Linked to Pelvic Endometriosis?
Brief Title: Organic Pollutants in Pelvic Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1072.6120.333.2021
Record Dates: First submitted 2023-03-05; First posted 2023-03-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Endometriosis; Infertility Unexplained
Keywords: Endometriosis, Unexplained Infertility, Polycyclic aromatic hydrocarbons
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: A prospective cohort tertiary-center study among women undergoing elective laparoscopy due to pelvic endometriosis (arm 1) or idiopathic infertility (arm 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endometriosis (Experimental): Women subjected to elective laparoscopy for pelvic endometriosis
  Interventions: Diagnostic Test: Detection of PAHs in visceral fat with gas chromatography-isotope dilution mass spectrometry
- idiopathic infertility (Active Comparator): Women subjected to elective laparoscopy for idiopathic infertility
  Interventions: Diagnostic Test: Detection of PAHs in visceral fat with gas chromatography-isotope dilution mass spectrometry

INTERVENTIONS:
Diagnostic Test: Detection of PAHs in visceral fat with gas chromatography-isotope dilution mass spectrometry — 1 ml sample of visceral fat collected during elective laparoscopy for detection of PAHS by gas chromatography-isotope dilution mass spectrometry

SUMMARY:
The health toxicity of polycyclic aromatic hydrocarbons (PAHs), present in air and food, generated during energy production and waste incineration, is well known. PAHs can activate the aryl hydrocarbon receptor, which may interact with classic estrogen receptors and modify estrogen-dependent inflammation in endometriosis. There is no data on the hypothetical role of PAHs in the etiopathogenesis of endometriosis. The aim was to compare PAHs concentrations in visceral fat in women with endometriosis and idiopathic infertility.

DETAILED DESCRIPTION:
A prospective cohort tertiary-center study includes women undergoing laparoscopy due to pelvic endometriosis (arm 1) or/and idiopathic infertility (arm 2). A sample of 1 ml of the greater omentum is collected intraoperatively for detection of 16 PAHs, i.e. acenaphthene, acenaphthylene, anthracene, fluoranthene, fluorene, naphthalene, phenanthrene, pyrene, benz[a]anthracene, benzo[b]fluoranthene, benzo[k]fluoranthene, benzo[ghi]perylene, benzo[a]pyrene, chrysene, dibenz[a,h]anthracene, and indeno[1,2,3-cd]pyrene, by gas chromatography-isotope dilution mass spectrometry method. The concentration of selected PAHs in visceral fat in both populations will be compared. The correlation of concentrations of selected PAHs with the occurrence of infertility, pelvic pain syndrome, intensity of pain, peritoneal adhesions and the degree of endometriosis will be checked.

ELIGIBILITY:
Inclusion Criteria:

i) age 18-45, ii) indications for surgical treatment of endometriosis, iii) indications for invasive diagnostics and surgical treatment of idiopathic infertility.

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Accumulation and detection of PAHs in women's visceral fat. | up to 6 months
  Detection and confirmation of the accumulation of PAHs (acenaphthene, acenaphthylene, anthracene, fluoranthene, fluorene, naphthalene, phenanthrene, pyrene, benz[a]anthracene, benzo[b]fluoranthene, benzo[k]fluoranthene, benzo[ghi]perylene, benzo[a]pyrene, chrysene, dibenz[a,h]anthracene, and indeno[1,2,3-cd]pyrene) in human adipose tissue by gas chromatography-isotope dilution mass spectrometry method.
Comparison of concentrations of 16 reference PAHs in women in both study arms. | up to 6 months
  Comparison of concentrations of 16 PAHs (acenaphthene, acenaphthylene, anthracene, fluoranthene, fluorene, naphthalene, phenanthrene, pyrene, benz[a]anthracene, benzo[b]fluoranthene, benzo[k]fluoranthene, benzo[ghi]perylene, benzo[a]pyrene, chrysene, dibenz[a,h]anthracene, and indeno[1,2,3-cd]pyrene) in both study arms using standard statistical methods.

SECONDARY OUTCOMES:
Evaluation of PAHs concentrations correlation with endometriosis degree | up to 6 months
  Assessment of 16 PAHs concentrations depending on the degree of endometriosis severity using standard statistical methods.
Evaluation of PAHs concentrations correlation with the intensity of pelvic pain | up to 6 months
  Assessment of 16 PAHs concentrations depending the intensity of pelvic pain in Numeric Rating Scale using standard statistical methods.
Evaluation of PAHs concentrations correlation with the presence and severity of peritoneal adhesions | up to 6 months
  Assessment of 16 PAHs concentrations depending on the presence and severity of peritoneal adhesions using standard statistical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Study Chair — Jagiellonian University; Iwona Gawron, Ph.D., Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland